CLINICAL TRIAL: NCT04720690
Title: Bioimpedence and Arterial Function Monitoring at Birth and in Infants: the BAMBI Study
Brief Title: Bioimpedence and Arterial Function Monitoring at Birth and in Infants
Acronym: BAMBI
Status: Recruiting | Type: Observational
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 20QC6217
Record Dates: First submitted 2021-01-08; First posted 2021-01-22 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Arterial Stiffness; Fetal Growth Retardation; Small for Gestational Age at Delivery; Pre-Eclampsia
MeSH Terms: conditions — Fetal Growth Retardation; Pre-Eclampsia | interventions — Pulse Wave Analysis; Stroke Volume; Cardiac Output; Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Appropriately grown for age infants: 40 appropriately grown for gestational age (AGA) infants. 20 will be <32 weeks, and 20 will be ≥32 weeks gestational age at birth.
  Interventions: Device: Vicorder: pulse wave velocity, pulse wave analysis, stroke volume, cardiac output; Device: NICaS; Device: Echocardiography and ultrasound of arteries
- Small for gestational age infants: 40 small for gestational age (SGA) infants. 20 will be <32 weeks, and 20 will be ≥32 weeks gestational age at birth.
  Interventions: Device: Vicorder: pulse wave velocity, pulse wave analysis, stroke volume, cardiac output; Device: NICaS; Device: Echocardiography and ultrasound of arteries
- Fetal growth restricted infants: 40 fetal growth restricted (FGR) infants. 20 will be <32 weeks, and 20 will be ≥32 weeks gestational age at birth.
  Interventions: Device: Vicorder: pulse wave velocity, pulse wave analysis, stroke volume, cardiac output; Device: NICaS; Device: Echocardiography and ultrasound of arteries

INTERVENTIONS:
Device: Vicorder: pulse wave velocity, pulse wave analysis, stroke volume, cardiac output — Measurement of arterial stiffness and cardiac output
Device: NICaS — Measurement of cardiac output
Device: Echocardiography and ultrasound of arteries — Measurement of cardiac output; measurement of intima-media thickness of arteries

SUMMARY:
Babies may be born appropriately grown for gestational age (AGA, >10th centile) or small for gestational age (SGA, <10th centile). Babies who are SGA and have evidence in utero of vascular compromise using antenatal doppler indices are classified as having fetal growth restriction (FGR). Babies with FGR are at increased risk of cardiovascular disease in adult life. Increased arterial stiffness and intima-media thickness are thought to mediate this risk in adults. It is not known how early in life these changes can be robustly detected. In addition, very little is known generally about how babies' hearts and arteries change in structure and function over the first year of life, whether affected by SGA or not. This study aims to understand if there are differences in cardiac and arterial structure and function between babies born AGA or SGA. Within the group of SGA babies, the study team will investigate whether FGR and maternal pre-eclampsia influence these measurements. The effects gestational age on these parameters will be studied within all groups: half of the babies recruited will be <32 weeks gestational age (GA), and half will be ≥32 weeks GA. Study participants will have further measurements at 3-6 months of life to assess if cardiac and arterial structure and function change in babies over the first year of life. The study team will use the Vicorder device to measure arterial stiffness, and assess the feasibility of using this device in neonates. The Vicorder will also be used to measure cardiac output. The feasibility and validity of this device for this purpose will be investigated (Vicorder is not validated for cardiac output measurement in infants). Vicorder cardiac output results will be compared to echocardiography and bioimpedence technology (using the NICaS monitor). The study team will use ultrasound for arterial structure measurements of the carotid artery and aorta.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term infants (including those with SGA+/-FGR) in the postnatal ward
* Term and Preterm infants (including those with SGA+/-FGR) admitted to the neonatal unit
* Written informed parental consent

Exclusion Criteria:

* Antenatal or postnatal diagnosis of complex/life-limiting congenital anomaly or genetic condition
* Infants with no realistic chance of survival
* Infants with fragile skin not permitting use of cuffs for research purposes
* Babies whose parents have a limited understanding of English will be excluded in the event that communication via NHS translation services is not possible due to clinical demands on these services

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All term and preterm infants born at the Imperial College Healthcare NHS trust can be included to the study after parental consent.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of arterial and cardiac function measurements: the proportion of babies from whom study measurements are successfully obtained. | 3 years
  Feasibility of arterial and cardiac function measurements assessed through establishing from what proportion of babies the team is able to successfully obtain these measurements.

SECONDARY OUTCOMES:
Non-invasive measurement of arterial stiffness: brachial-femoral pulse wave velocity | 3 years
  Brachial-femoral pulse wave velocity in metres per second (m/s) will be measured using the Vicorder and compared between neonates of different gestational age and birth weight groups at or near term corrected gestational age, and at 3-6 months of age.
Non-invasive measurement of arterial stiffness: augmentation index | 3 years
  Augmentation index (%) will be measured using the Vicorder and compared between neonates of different gestational age and birth weight groups at or near term corrected gestational age, and at 3-6 months of age.
Arterial structure measurements | 3 years
  The intima-media thickness of the carotid artery and abdominal aorta will be measured in micrometres (µm) using ultrasound at or near term corrected gestational age, and at 3-6 months of age. Gestational age and birth weight groups will be compared at each time point.
Cardiac output measurements: comparison of neonatal and infant birth weight and gestational age cohorts | 3 years
  Cardiac output in L/min and ml/min/kg will be measured using echocardiography, the NICaS monitor and the Vicorder. Values obtained in different gestational age and birth weight groups will be compared at or near term corrected gestational age and at 3-6 months of age.
Cardiac output measurements: comparison of devices | 3 years
  Cardiac output values in L/min and ml/min/kg obtained by each device (echocardiography, NICaS monitor and Vicorder) will be compared using correlation and Bland-Altman statistics.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Queen Charlotte's and Chelsea Hospital, London
  - St Mary's Hospital, London

IPD SHARING:
Plan to Share IPD: No